CLINICAL TRIAL: NCT05824754
Title: Pilot Project 1. Feasibility Pilot of a JITAI to Reduce Cannabis Use Among Emerging Adults
Brief Title: An App to Reduce Cannabis Use Among Emerging Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Inbal Billie Nahum-Shani, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00222194; 5P50DA054039-02 (NIH)
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cannabis Use
Keywords: Cannabis Use; Marijuana; Substance-Related Disorders; Mental Disorders
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JITAI (Experimental): Experimental: Within-participant micro-randomization
  Twice daily in the study, a participant is assigned to receive a message or no message. The micro-randomization will be performed by a reinforcement learning algorithm based on the participant's engagement with the intervention.
  Interventions: Other: Just-In-Time-Adaptive-Intervention (JITAI)

INTERVENTIONS:
Other: Just-In-Time-Adaptive-Intervention (JITAI) — Behavioral: MiWaves behavioral messages
  Participants will be using the MiWaves mobile app for 30 days. When a participant is assigned to receive a message, a message will be randomly selected from a pool of intervention message sets. Messages are based in motivational interviewing and include affect management and behavioral economic strategies.

SUMMARY:
This study is being completed to pilot prevention methods to promote wellness and reduce risky behaviors, including the use of substances such as cannabis. This study will help researchers learn about ways of delivering this information that is both appealing and helpful to young adults who use mobile apps.

ELIGIBILITY:
Inclusion Criteria:

* Reside in the US
* Speak and read English
* Have a smartphone on which the app can be downloaded
* Screen positive for cannabis use 3 or more times each week over the past month
* Report motivation to change cannabis as 1 or higher (using scale of 0-10)
* Meet Study verification criteria (i.e., use of CAPTCHA, IP address checks)

Exclusion Criteria:

* Use of Medical Cannabis
* Failure to meet study verification criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- JITAI: Experimental: Within-participant micro-randomization
  Twice daily in the study, a participant is assigned to receive a message or no message. The micro-randomization will be performed by a reinforcement learning algorithm based on the participant's engagement with the intervention.
  Just-In-Time-Adaptive-Intervention (JITAI): Behavioral: MiWaves behavioral messages
  Participants will be using the MiWaves mobile app for 30 days. When a participant is assigned to receive a message, a message will be randomly selected from a pool of intervention message sets. Messages are based in motivational interviewing and include affect management and behavioral economic strategies.
Period: Overall Study
Arm/Group | JITAI
Started | 122
Completed | 122
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | JITAI
Number analyzed (Participants) | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 115
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 89
  More than one race | 14
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 122

OUTCOME MEASURES:

1. Primary Outcome: App Feasibility
Description: % of participants who consented to the study who download the MiWaves app.
Time Frame: 1 month
Population: App feasibility outcome is operationalized as % of participants who consented to the study who download the MiWaves app. Not all that consented to the study were included in study flow since not all that consented downloaded the app. Therefore, the number analyzed for app feasibility is greater than the number in the participant flow.
Measure: Count of Participants; unit: Participants
Arm/Group | JITAI
Number analyzed (Participants) | 137
Participants | 122

2. Primary Outcome: App Acceptability
Description: Participants will complete acceptability ratings for the MiWaves app within their post-test assessment (percent with positive rating).
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | JITAI
Number analyzed (Participants) | 112
Participants | 90

ADVERSE EVENTS:
Time Frame: Up to 2.5 months. After enrollment, participants were followed for AEs until either: a) The participant completes the follow-up survey (2-months post enrollment) b) The window for completing the follow-up survey passed (2 weeks after sending follow-up survey) Therefore, the maximum amount of time a participant would be followed for AEs is 2.5 months post-enrollment.
Description: There are no adverse events to report.
Arm/Group | JITAI
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 0/122
Other Adverse Events (participants affected / at risk) | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT05824754/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT05824754/ICF_001.pdf